CLINICAL TRIAL: NCT03661476
Title: Investigation of the Effect of Oculo-Motor Exercises in Intermittent Exotropic Children
Brief Title: The Effect of Oculo-Motor Exercises in Intermittent Exotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, PhD PT, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.34141
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-03

CONDITIONS: Intermittent Exotropia; Exercises
Keywords: Intermittent Exotropia; Oculo-Motor Exercises; Physiotherapy; Intermittent Exotropia Survey
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oculo-Motor Exercises (OME) (Experimental): 10 repetitive four different oculomotor exercise protocols with eye stabilization were organized as home programs for 6 weeks, twice a day in the morning and evening each day of the week.
  Interventions: Behavioral: Oculo-Motor Exercises (OME)

INTERVENTIONS:
Behavioral: Oculo-Motor Exercises (OME) — Oculomotor Exercises (OME); The saccadic eye movement exercise included moving the eyes horizontally between two stationary targets while keeping the head still.
  The smooth pursuit exercise included moving the target horizontally and tracking it with the eyes while keeping the head still.
  The adaptation X1 exercise included moving the head horizontally while keeping the stationary target in focus.
  The adaptation X2 exercise included moving the head and target in opposite directions horizontally while tracking the target with the eyes.

SUMMARY:
In childhood strabismus, exotropia is most frequently seen with intermittent exotropia and convergence failure in the first decade of life. This situation adversely affects children's psychosocial development and creates worries about personal relationships and work life in their future lives. Patients' hesitant attitudes towards surgical treatment led to the out-of-surgery techniques such as exercise therapy. No studies have been found in the literature on the efficancy of the intermittent exotropia treatments with oculo-motor exercises. In our study, it was aimed to investigate the effects of oculo-motor exercises on intermittent exotropia in children.

DETAILED DESCRIPTION:
50 volunteer school-aged children between 2-17 years of age) were included in our study. Oculo-motor home exercise protocols were given to all participants for 2 sessions per day for 6 weeks, and regular phone calls were made once a week. Participants were assessed cycloplegic refraction by autorefractometry, corrected and uncorrected visual acuity by snellen chart, ocular motility test, near and distant alternating prism cover test, streopsis test and patient satisfaction levels by intermittent exotropia survery.

ELIGIBILITY:
Inclusion Criteria:

* Be between 2 and 17 years of age
* Intermittent exotropia diagnosis
* To have mental capacity in the level to understand and do exercises

Exclusion Criteria:

* Not complying with age criteria
* Constant exotropia
* Having undergone eye surgery
* Those with systemic disease that prevent exercise

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Prism cover test | 6 weeks
  Near and distant alternating prism cover test

SECONDARY OUTCOMES:
Streopsis test | 6 weeks
  Three-dimensional visual assessment
Intermittent exotropia survery | 6 weeks
  Level of patient satisfaction
Visual acuity | 6 weeks
  Snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Candan Algun, Study Director — Faculty of Health Sciences
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Govindan M, Mohney BG, Diehl NN, Burke JP. Incidence and types of childhood exotropia: a population-based study. Ophthalmology. 2005 Jan;112(1):104-8. doi: 10.1016/j.ophtha.2004.07.033. PMID 15629828
- [Result] Joyce KE, Beyer F, Thomson RG, Clarke MP. A systematic review of the effectiveness of treatments in altering the natural history of intermittent exotropia. Br J Ophthalmol. 2015 Apr;99(4):440-50. doi: 10.1136/bjophthalmol-2013-304627. Epub 2014 Jul 7. PMID 25001323
- [Result] Morimoto H, Asai Y, Johnson EG, Lohman EB, Khoo K, Mizutani Y, Mizutani T. Effect of oculo-motor and gaze stability exercises on postural stability and dynamic visual acuity in healthy young adults. Gait Posture. 2011 Apr;33(4):600-3. doi: 10.1016/j.gaitpost.2011.01.016. Epub 2011 Feb 19. PMID 21334899